CLINICAL TRIAL: NCT02283307
Title: Dual Energy CT Urography Using 50% Reduction in Iodinated Contrast: Feasibility, Image Quality, and Radiation Dose Reduction With Virtual Unenhanced Images.
Brief Title: Dual Energy CT Urography With Reduced Iodinated Contrast
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Responsible Party: Principal Investigator, William Shuman, Professor and Vice Chair of Radiology, University of Washington
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 47637
Record Dates: First submitted 2014-10-09; First posted 2014-11-05 (Estimated); Last update posted 2018-05-14 (Actual); Status verified 2018-05

CONDITIONS: Aortic Aneurysm
MeSH Terms: conditions — Aortic Aneurysm

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Reduced contrast DECT scan (Experimental): Reduced Contrast Dual Energy CT
  Interventions: Other: Reduced contrast DECT scan; Other: Standard contrast SECT scan

INTERVENTIONS:
Other: Reduced contrast DECT scan — Subjects will undergo a dual energy CT scan with reduced contrast
Other: Standard contrast SECT scan — Subjects will undergo standard of care single energy CT scan with a standard dose of contrast. (control)

SUMMARY:
The goal of this study is to validate that Dual Energy CT (DECT) urography when performed with a 50% reduction in iodinated contrast dose results in a CT exam with equal or better image quality and equal or better diagnostic capability compared to traditional Single Energy CT (SECT) performed with a standard contrast dose.

DETAILED DESCRIPTION:
The investigators hypothesize that DECT urography performed with a 50% iodine dose reduction is equivalent to SECT urography performed with a full iodine dose for:

* Enhancement of the aorta, renal arteries, and renal veins
* Enhancement of the renal cortex
* Enhancement of the renal pelvis, ureters, and bladder
* Subjective evaluation of image quality
* Objective evaluation of image quality

In addition, the investigators hypothesize that DECT virtual non-contrast images using material suppression from the same low iodine CT exam results in equivalent diagnostic information compared to SECT true non-contrast images obtained in the same patient during the same exam. If the true non-contrast images could be replaced by the virtual non-contrast images without loss of information, there is potential for DECT to both significantly lower radiation dose as well as significantly decreasing iodine dose.

The investigators designed this research protocol to prospectively test these hypotheses in a population scanned with a 50% reduced iodine DECT urography protocol compared to a control population scanned with a standard iodine dose clinical SECT urography protocol.

ELIGIBILITY:
Inclusion Criteria:

* Age >50
* Outpatient scheduled to have a CT urography at the site

Exclusion Criteria:

* Severe allergy to iodine containing contrast
* Pregnancy (which is very unlikely for those over 50)
* Body mass index (BMI) over 35 kg/m2
* Inability to provide informed consent
* Inpatient

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2014-09; Primary Completion 2017-08 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Diagnostic ability determined by image quality (subjective and objective evaluation of vessel attenuation and depiction, image noise, image quality and information from virtual non-contrast | Up to 24 months

CONTACTS AND LOCATIONS:
Locations (1):
- University of Washington Medical Center, Seattle, Washington, United States